CLINICAL TRIAL: NCT07198984
Title: Isolate and Characterise Probiotics Capable of Increasing Butyrate Production in Order to Develop Products That Improve Gut Health and Microbiota Balance
Brief Title: Boosting Microbiota Butyrate Producers to Improve Gut Health
Acronym: BOOST-Mi
Status: Recruiting | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00623-46
Record Dates: First submitted 2025-09-12; First posted 2025-09-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Adults 20 to 80 Years

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The human gut microbiota is a dynamic ecosystem essential to health, influenced by diet, age, and lifestyle. It plays a key role in digestion, immunity, and nervous system regulation. Among its important compounds, short-chain fatty acids, particularly butyrate, are crucial for intestinal and metabolic balance, as they support homeostasis, strengthen the epithelial barrier, and have anti-inflammatory effects.

An imbalance in the microbiota, especially a decrease in butyrate-producing bacteria, is linked to intestinal, metabolic, and neurological disorders. A fiber-rich diet promotes the growth of these beneficial bacteria.

This study aims to isolate and characterize probiotics that can enhance butyrate production, thereby improving intestinal health and microbiota balance. Sampling conditions will comply with regulations governing research involving human subjects.

DETAILED DESCRIPTION:
The human gut microbiota is a complex and adaptable ecosystem closely linked to its host, influenced by factors such as diet, lifestyle, and age. It plays key roles in nutrition, immunity, and pathogen protection by breaking down otherwise indigestible fibers into short-chain fatty acids, which are essential for energy production, metabolism, and immune balance.

Butyrate, the best-studied short-chain fatty acids, provides most of the energy for colonic cells, strengthens the intestinal barrier, reduces inflammation, and regulates gene expression related to cell growth, apoptosis, and autophagy. A decrease in butyrate-producing bacteria has been associated with intestinal, metabolic, neurological, and other diseases, including rheumatoid arthritis and fatty liver disease.

Maintaining a healthy microbiota-particularly through a fiber-rich diet that supports butyrate producers-is essential for digestion, nutrient absorption, immune regulation, and overall health, highlighting the strategic role of butyrate in disease prevention and well-being.

This project hypothesizes that increasing microbiota-derived butyrate could improve gut health. Its aim is to isolate and characterize probiotic strains capable of boosting butyrate production, in order to develop scientifically grounded, high-functionality probiotic products. The study will also assess whether butyrate production correlates with beneficial in vitro effects and further clarify how butyrate producers interact with both the microbiota and the host.

ELIGIBILITY:
Inclusion Criteria:

* People between the ages of 20 and 80, in good health, with a body mass index between 18.5 kg/m² and 30 kg/m², who are not deprived of their liberty or under guardianship.
* Additional criteria for people aged between 20 and 60: Engaging in sports at least twice a week or following a flexitarian diet, No known chronic conditions, Not undergoing chronic treatment.

Exclusion Criteria:

* Under the age of 20 or over the age of 80, Part of the principal investigator's team, Reporting to the investigator (intern, student, or employee under their authority), Having been on antibiotic therapy in the 3 months prior to sampling, Having taken probiotics in the 15 days prior to sampling, Having taken synbiotics in the 15 days prior to sampling, Having a BMI below 18.5 kg/m² or above 30 kg/m², Being deprived of liberty or under guardianship.
* Additional criteria for people aged between 20 and 60: Not exercising twice a week or following a flexitarian diet, Having a chronic illness, Undergoing chronic treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of bacterial strains identified from stool samples that belong to species known to produce butyrate or stimulate butyrate production (16S rRNA gene sequencing) | up to 3 years
  Stool samples will be collected from participants and processed under anaerobic conditions to maximize bacterial survival. Homogenized samples will be plated on selective culture media and incubated at 37 °C under aerobic or anaerobic conditions. Clones will be expanded in liquid culture, and isolated bacterial strains will be identified by 16S rRNA gene sequencing. The outcome will be reported as the number of distinct strains belonging to species with documented butyrate-producing capacity. The primary endpoint is the identification of at least 12 such strains.

CONTACTS AND LOCATIONS:
Locations (1):
- INRAE, Jouy-en-Josas, France

IPD SHARING:
Plan to Share IPD: No